CLINICAL TRIAL: NCT01213173
Title: A Randomised, Open Label, Parallel Group, Multicentre, Phase IV Study on the Effect of 8 Weeks Succinate Metoprolol (Betaloc ZOK®) (95 - 190 mg) on Heart Rate in the Stable Angina Patients
Brief Title: Evaluation of Succinate Metoprolol on Heart Rate in the Stable Angina Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4022L00008
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Results first posted 2013-08-26 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Angina Pectoris
Keywords: angina pectoris; chest pain; heart rate
MeSH Terms: conditions — Angina Pectoris; Chest Pain | interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Succinate Metoprolol (Betaloc ZOK®)
- 2 (Experimental)
  Interventions: Drug: Succinate Metoprolol (Betaloc ZOK®)

INTERVENTIONS:
Drug: Succinate Metoprolol (Betaloc ZOK®) — treatment with 47.5mg for two weeks, if tolerated and without Systolic blood pressure<100mmHg and heart rate <45 bpm according to 12-lead Electrocardiogram at Week 3, the dosage will be titrated to 95mg and last for another 6 weeks
  Arms: 1
Drug: Succinate Metoprolol (Betaloc ZOK®) — Treatment with 95mg for two weeks, and if tolerated and without bradycardia symptoms presented, Systolic blood pressure<100mmHg and heart rate <45 bpm according to 12-lead Electrocardiogram at Week 3，the dosage will be force titrated to 190mg and last for another 6 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effects of Succinate Metoprolol(Betaloc ZOK®) (95 - 190 mg) on heart rate in the Stable angina patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Chinese patients
* Heart rate ≥ 65bpm
* Has been diagnosed as Stable angina for at least 1 month and with stable angina pectoris symptoms within 2 weeks previous to enrolment(Please find the diagnose criteria of Stable angina on Appendix C)
* With Left ventricular ejection fraction ≥ 50% according to ultrasound cardiogram;
* Has been on beta-blockers for at least 4 weeks*, on the dose equivalent to Betaloc ZOK® 23.75-47.5mg/day.

Exclusion Criteria:

* Acute myocardial infarction within 6 months
* Unstable angina or Prinzmetal's angina
* II degree of AV block or greater
* Significant clinical, laboratory or electrocardiographic abnormalities that would place the subject at undue risk (in the Investigator's opinion) including:
* Significant renal impairment (serum creatinine > 2.0 mg/dL)
* Serum Alanine Aminotransferase or Aspartate Aminotransferase > 3 x upper limit of reference range
* Serum potassium < 3.0 mEq/L
* Serum sodium ≤ 130 mEq/L
* Acute or chronic hepatitis or cirrhosis (clinical diagnosis)
* Uncontrolled hyperthyroidism (clinical diagnosis)
* Systolic blood pressure ≥ 180 mmHg, or < 100mmHg at enrolment
* Patients with unstable, not compensated heart failure (pulmonary oedema, hypoperfusion or hypotension)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huo Yong, Principal Investigator — Department of Cardiology, Peking University First Hospital; Helen Lin, Study Director — Astrazeneca China
Locations (10):
- China (10):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Tangshan, Hebei
  - Research Site, Zhengzhou, Henan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Jingzhou, Liaoning
  - Research Site, Shenyang, Liaoning
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Tianjing

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=331&filename=CSR-D4022L00008.pdf
- See also: CSR-D4022L00008.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=331&filename=CSR-D4022L00008.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety Population is divided according to the actual dosage received by the patient, not the randomization. The patient will be high-dose group if the highest dose ever used is above 95mg; otherwise (if the highest dose ever used is equal to or lower than 95 mg) he/she will be low-dose group.
Pre-assignment Details: Safety population- patients who received at least 1 dose of investigational product. During initial 1 week run-in period subjects were treated with 47.5mg Betaloc ZOK®. Patients started to take investigational product before randomization therefore, number of subjects in Safety population (274) is greater than number of randomized and treated (251)
Groups:
- Active Comparator: lead Electrocardiogram at Week 3, the dosage will be titrated to 95mg and last for another 6 weeks
- Experimental: lead Electrocardiogram at Week 3，the dosage will be force titrated to 190mg and last for another 6 weeks
Period: Overall Study
Arm/Group | Active Comparator | Experimental
Started | 125 (Patients who were randomized and received treatment) | 126 (Patients who were randomized and received treatment)
Patients Included in Safety Population | 139 | 112
Patients Included in ITT Population | 116 | 115
Patients Included in PP Population | 102 | 89
Completed | 113 (Patients who completed the study) | 110 (Patients who completed the study)
Not Completed | 12 | 16
Not completed — Protocol Violation | 2 | 0
Not completed — Adverse Event | 4 | 8
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Incorrect Enrollment | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator | Experimental | Total
Number analyzed (Participants) | 116 | 115 | 231
Age, Continuous [Mean (Standard Deviation); unit: Year] | 59.3 (7.81) | 59.2 (9.25) | 59.2 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 81 | 155
  Male | 42 | 34 | 76

OUTCOME MEASURES:

1. Primary Outcome: The Impact on 24-hr Average Heart Rate Between Two Groups (Betaloc ZOK® 95mg vs. 190mg)
Description: Difference of the 24-hr average heart rate between two groups after 8 weeks treatment.
Time Frame: After 8 weeks treatment in the study
Population: ITT population was defined as all randomized subjects who had taken at least one dose of trial treatment, who had measurements at baseline for one or more efficacy variables and at least one post baseline measurement for the same variables in the treatment period.
Measure: Mean (Standard Deviation); unit: Bpm
Groups:
- Arm 1 - Active Comparator: Drug: Succinate Metoprolol (Betaloc ZOK®) Treatment with 47.5mg for two weeks, if tolerated and without Systolic blood pressure<100mmHg and heart rate <45 bpm according to 12-lead Electrocardiogram at Week 3, the dosage will be titrated to 95mg and last for another 6 weeks
- Arm 2 - Experimental: Drug: Succinate Metoprolol (Betaloc ZOK®) Treatment with 95mg for two weeks, and if tolerated and without bradycardia symptoms presented, Systolic blood pressure<100mmHg and heart rate <45 bpm according to 12-lead Electrocardiogram at Week 3，the dosage will be force titrated to 190mg and last for another 6 weeks
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 116 | 115
Bpm
  Baseline | 71.4 (8.02) | 70.9 (8.19)
  Week 9 | 70.9 (8.71) | 68.6 (8.40)

2. Secondary Outcome: The Impact on 24-hr Average Heart Rate From Baseline Within Groups
Description: Difference of the 24-hr average heart rate within groups from baseline after 8 weeks treatment.
Time Frame: After 8 weeks treatment in the study
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Bpm
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 116 | 115
Bpm | -0.6244 (7.16) [-1.94 to 0.69] | -2.9858 (6.62) [-4.23 to -1.75]

3. Secondary Outcome: The Different Impact on 24-hr Average Heart Rate Between Two Groups
Description: Difference of the 24-hr average heart rate between two groups after 2 weeks of treatment.
Time Frame: After 2 weeks treatment in the study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Bpm
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 116 | 115
Bpm | 70.6 (7.75) | 69.2 (7.82)

4. Secondary Outcome: The Different Impact on 24-hr Average Heart Rate From Baseline Within Groups
Description: Difference of the 24-hr average heart rate within groups from baseline after 2 weeks treatment.
Time Frame: After 2 weeks treatment in the study
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Bpm
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 116 | 115
Bpm | -0.4938 (4.69) [-1.40 to 0.41] | -2.1383 (5.71) [-3.18 to -1.10]

5. Secondary Outcome: The Proportion of Patients With Resting Heart Rate Controlled to ≤60bpm Between Groups
Description: Difference in proportions of patients who had resting heart rate controlled to ≤60 bpm after 2 weeks treatment between groups
Time Frame: After 2 weeks treatment
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 116 | 115
Participants | 25 | 28

6. Secondary Outcome: The Proportion of Patients With Resting Heart Rate Controlled to ≤60bpm Between Groups
Description: Difference in proportions of patients who had resting heart rate controlled to ≤60 bpm after 8 weeks treatment between groups
Time Frame: After 8 weeks treatment
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 116 | 115
Participants | 28 | 46

7. Secondary Outcome: The Difference of Change From Baseline in Total Ischemic Burden Between Groups
Description: Difference in change from baseline in TIB between two groups after 2 weeks treatment.
  Total Ischemic Burden (TIB) was defined as the sum of product of each ischemia episode lasting time and maximal ST elevation: TIB=Σ(STmax×Tisc).
Time Frame: After 2 weeks treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm*min
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 116 | 115
mm*min | -5.3353 (69.0874) [-15.1422 to 4.4716] | -12.9874 (66.3041) [-20.8416 to 5.1332]

8. Secondary Outcome: The Difference of Change From Baseline in Total Ischemic Burden Between Groups
Description: Difference in change from baseline in TIB between two groups after 8 weeks treatment.
  Total Ischemic Burden (TIB) was defined as the sum of product of each ischemia episode lasting time and maximal ST elevation: TIB=Σ(STmax×Tisc).
Time Frame: After 8 weeks treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm*min
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 116 | 115
mm*min | 22.2905 (112.1215) [-14.3181 to 58.8992] | -7.6586 (79.1887) [-18.6777 to 3.3604]

9. Secondary Outcome: The Difference of Change From Baseline in Angina Frequency Between Groups
Description: Difference in change from baseline of angina pectoris frequency between two groups after 2 weeks treatment.
Time Frame: After 2 weeks treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Attacks per week
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 116 | 115
Attacks per week | -0.044 [-0.40 to 0.31] | -0.3243 [-0.55 to -0.10]

10. Secondary Outcome: The Difference of Change From Baseline in Angina Frequency Between Groups
Description: Difference in change from baseline of angina pectoris frequency between two groups after 8 weeks treatment.
Time Frame: After 8 weeks treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Attacks per week
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 116 | 115
Attacks per week | -0.3930 [-0.64 to -0.14] | -0.4453 [-0.71 to -0.18]

11. Secondary Outcome: The Change From Baseline in Total Cholesterol
Description: Difference of change from baseline in TC after 8 weeks treatment between groups.
Time Frame: After 8 weeks treatment
Population: All subjects who received at least one dose of randomized investigational product was included in the safety population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 139 | 112
mmol/L | -0.0505 (0.8949) [-0.7110 to 0.6101] | 0.5825 (4.6175) [-0.1029 to 1.2678]

12. Secondary Outcome: The Change From Baseline in Fasting Plasma Glucose
Description: Difference of change from baseline in FPG after 8 weeks treatment between groups.
Time Frame: After 8 weeks treatment
Population: All subjects who received at least one dose of randomized investigational product was included in the safety population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 139 | 112
mmol/L | 0.3844 (1.7130) [-0.1127 to 0.6560] | 0.2487 (0.8809) [-0.0344 to 0.5318]

13. Secondary Outcome: The Change From Baseline in Triglycerides
Description: Difference of change from baseline in TG after 8 weeks treatment between groups.
Time Frame: After 8 weeks treatment
Population: All subjects who received at least one dose of randomized investigational product was included in the safety population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Arm 1 - Active Comparator | Arm 2 - Experimental
Number analyzed (Participants) | 139 | 112
mmol/L | 0.1295 (0.7607) [-0.0375 to 0.2965] | 0.0937 (1.1520) [-0.0810 to 0.2683]

ADVERSE EVENTS:
Arm/Group | Active Comparator | Experimental
Serious Adverse Events (participants affected / at risk) | 1/139 | 3/112
Other Adverse Events (participants affected / at risk) | 0/139 | 0/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator (N=139) | Experimental (N=112)
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Genital neoplasm malignant female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0
angina unstable (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The sample size was insufficient for the secondary endpoints. Besides, the treatment prior to study did not correlate well with 47.5 mg metoprolol succinate, but with some higher dose. last the quality control of the study needs further improvement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less